CLINICAL TRIAL: NCT03655756
Title: Phase 1 Study Using a Plasmid DNA Coding for Emm55 Streptococcal Antigen in Patients With Unresectable Stage III or Stage IV Cutaneous Melanoma
Brief Title: pDNA Intralesional Cancer Vaccine for Cutaneous Melanoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: TuHURA Biosciences, Inc. (Industry)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM 2017-01
Record Dates: First submitted 2018-08-23; First posted 2018-08-31 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Cutaneous Melanoma, Stage III; Cutaneous Melanoma, Stage IV
Keywords: Unresectable; Melanoma; pDNA; Plasmid DNA; Gene Therapy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IFx-Hu2.0 (plasmid DNA) 0.1 mg/lesion/time point (Experimental): Therapeutic Classification:
  * Noncellular, Therapeutic Cancer Vaccine > Immunomodulator
  Route of Administration:
  * Intratumoral injection of cutaneous, subcutaneous or nodal lesions
  Mechanism of Action:
  * Injection of the IFx-Hu2.0 plasmid DNA construct into the target lesion facilitates the localized expression of the highly immunogenic Emm55 protein by the tumor cells on their cell surface.
  Physiological Effect:
  * This expression then primes a cascade of immune events that exposes the patient-specific abnormal tumor antigens to the effector mechanisms of the immune system. The immune response becomes systemic as inter-antigenic epitope spreading produces neoantigens to naïve T cells. Therefore, injected lesions are targeted along with non-injected lesions (abscopal effect). This is especially important in conditions where the mutational phenotype varies greatly among individual lesions.
  Interventions: Biological: IFx-Hu2.0

INTERVENTIONS:
Biological: IFx-Hu2.0 — Subjects enrolled will receive a fixed IFx-Hu2.0 (plasmid DNA) dose of 0.1 mg injected in up to 3 lesions at a single time point (28-day follow-up post last injection).
  Other Names: pAc/emm55

SUMMARY:
Six patients will receive IFx-Hu2.0 on an outpatient basis at a single time point in a single lesion, two lesions, or three lesions, as a monotherapy (a maximum of three lesions could be injected). These patients will be assessed for any immediate adverse reactions and at Week 4 (Day 28+/-7 business days for any delayed adverse events.

DETAILED DESCRIPTION:
Six male and/or female adult patients (greater than or equal to 18 years old), of any ethnicity and race, with unresectable stage III or stage IV cutaneous melanoma with accessible lesions, will be eligible for enrollment and treatment with IFx-Hu2.0.

To be eligible for this study, patients with unresectable metastatic disease must have failed, refused or been deemed not candidates for at least one form of systemic anti-PD-1-based immunotherapy as well as BRAF inhibition, if BRAF V600 mutated. Talimogene laherparepvec (IMLYGIC®) is indicated for local treatment of unresectable cutaneous, subcutaneous, and nodal lesions in patients with melanoma recurrent after initial surgery. Therefore, patients with unresectable cutaneous, subcutaneous, and nodal melanoma lesions recurrent after initial surgery must have failed, refused or been deemed not candidates for talimogene laherparepvec to be eligible for this study.

Enrollees will receive IFx-Hu2.0 at a single time point. Depending on the number of accessible lesions, a patient could receive up to three doses across three lesions (one dose per lesion). Forty milliliters of peripheral blood will be collected from these patients prior to treatment administration and at the follow-up visit four weeks later. The target dose will be 100 μg of plasmid DNA per lesion injected at a final dose volume of 200 μL per lesion. To allow for the observation of any acute toxicity in the first subject enrolled and prevent any occurrence of excessive toxicities in subsequent subjects, the first subject enrolled will receive a single dose of IFx-Hu2.0. Subsequent subjects will be administered the product after at least seven days. Beyond the first subject, the maximum number of lesions to be injected at any given time point in the study phase proposed is three lesions. These samples will be used to perform complete blood counts (CBC) and clinical chemistry tests. A urine sample will be obtained for urinalysis for protein and blood at the same frequency. Blood samples will be drawn for immune response evaluation as well. At the end of the study period, a biopsy of the lesion injected and a non-injected lesion (if applicable) will be collected. If the patient has a response to therapy, the patient will have the option of continuing the study at three-week intervals so long as they have not progressed. Optional tumor biopsies and peripheral blood collections may be obtained on subsequent treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable stage III or stage IV malignant melanoma, with accessible cutaneous lesions
* Must have measurable disease greater than 3 mm
* At least one injectable lesion and one lesion for biopsy at study conclusion. Lymphocyte count ≥ 500,000 cells/mL
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Willing and able to give written, informed consent
* If male or female of childbearing potential must be willing to use a contraceptive during the study and for six months afterward. A woman is considered to be of childbearing potential unless she has had a surgical procedure that would accomplish sterility such a bilateral tubal ligation, hysterectomy or has not had menses for the past 12 months.
* Life expectancy greater than three months
* To be eligible for this study, patients with unresectable metastatic disease must have failed, refused or been deemed not candidates for at least one form of systemic anti-PD-1-based immunotherapy as well as BRAF inhibition, if BRAF V600 mutated.
* Patients with unresectable cutaneous, subcutaneous, and nodal melanoma lesions recurrent after initial surgery must have failed, refused or been deemed not candidates for talimogene laherparepvec to be eligible for this study.
* The entry laboratory criteria for subject eligibility must be less than or equal to grade 1 adverse event levels for the parameters tested as defined by CTCAE v5.0.

Exclusion Criteria:

* Known brain metastases greater than 1 cm at screening.
* Life expectancy of fewer than three months
* Prior systemic anti-cancer treatment within three weeks from start of treatment (Day 0)
* Current treatment with systemic immunosuppressive corticosteroid (greater than 10 mg of daily prednisone) doses or other immunosuppressants such as those needed for solid organ transplants. Medications needed to treat conditions such as reactive airway disease are not excluded.
* Pregnant or lactating women
* Presence of any uncontrolled and significant medical or psychiatric condition which would interfere with trial safety assessments
* Treatment with any investigational product within the three weeks preceding injection
* Immunizations for encapsulated bacteria were not given for patients who have undergone a splenectomy.
* Serious underlying medical or psychiatric conditions, active infections requiring the use of antimicrobial drugs, or active bleeding that would make the subject unsuitable or unable to participate in the study
* Concurrent chemotherapy or biological therapy. Concurrent radiotherapy is allowed as long as it is not the same site as the injected lesion.
* Uncontrolled hepatitis B, hepatitis C, or HIV infection
* History of organ allograft transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Markowitz, MD, PhD, Principal Investigator — Collaborator
Locations (1):
- H. Lee Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had a goal of six evaluable patients. It was the intent of the study team to recruit an additional two patients to be screened and enrolled if any of the existing patients were lost to follow-up, withdrew consent, or exhibited disease progression.
Groups:
- IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion/Time Point: Therapeutic Classification:
  * Noncellular, Therapeutic Cancer Vaccine > Immunomodulator
  Route of Administration:
  * Intratumoral injection of cutaneous, subcutaneous or nodal lesions
  Mechanism of Action:
  * Injection of the IFx-Hu2.0 plasmid DNA construct into the target lesion facilitates the localized expression of the highly immunogenic Emm55 protein by the tumor cells on their cell surface.
  Physiological Effect:
  * This expression then primes a cascade of immune events that exposes the patient-specific abnormal tumor antigens to the effector mechanisms of the immune system. The immune response becomes systemic as inter-antigenic epitope spreading produces neoantigens to naïve T cells. Therefore, injected lesions are targeted along with non-injected lesions (abscopal effect). This is especially important in conditions where the mutational phenotype varies greatly among individual lesions.
  IFx-Hu2.0: Subjects enrolled will receive a fixed IFx-Hu2.0 (plasmid DNA) dose of 0.1 mg injected in up to 3 lesions at a single time point (28-day follow-up post last injection).
Period: Overall Study
Arm/Group | IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion/Time Point
Started | 7
Completed | 6
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion/Time Point
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
AJCC Clinical Staging [Count of Participants; unit: Participants] — Stage III: tumor no more than 2mm thick and could be ulcerated. Cancer has spread to 1-3 nearby nodes. It has not spread to distant parts of the body.
  Stage IIIC: tumor no more than 2mm thick with 1-3 macroscopic node metastases and an ulcerated primary melanoma. Patients with satellite(s)/in-transit metastases, or any patient with nodal disease regardless of ulceration status.
  Stage IV: tumor of any thickness and could be ulcerated. Cancer could have spread to nearby nodes. It has spread to distant nodes or to organs.
  Note: lesser stages correlate with improved outcomes.
  Participants
    Stage III | 1
    Stage III C | 4
    Stage IV | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and/or Dose Limiting Toxicities (DLTs)
Description: Safety was reported using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Feasibility was defined as the ability to treat at least five of the six patients enrolled without drug-related dose-limiting toxicity (DLT).
Time Frame: 28 ± 7 Days
Population: The data analysis is described to assess the safety of the injection of the study agent in six patients the intention-to-treat (ITT) approach will be used for response to treatment data analysis of this trial (secondary objective).
Measure: Count of Participants; unit: Participants
Arm/Group | IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion/Time Point
Number analyzed (Participants) | 6
Participants
  Participants Analyzed | 6
  Serious Adverse Events (SAEs) | 1
  Dose Limiting Toxicity (DLT) | 0

2. Secondary Outcome: Antitumor Response Induced by IFx-Hu2.0 Per RECIST v1.1 for Target Lesions.
Description: Evaluation of response rate and assessment of the antitumor immune responses induced by IFx-Hu2.0 per RECIST v1.1 for target lesions.
  Complete Response (CR), Disappearance of all target lesions. Partial Response (PR), ≥ 30% decrease in the sum of the longest diameters of target lesions compared with baseline.
  Stable Disease (SD), Neither sufficient shrinkage to qualify for partial or complete response (CR or PR) nor sufficient increase to qualify for progressive disease (PD).
  Progressive Disease (PD), Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 28 ± 7 days post treatment
Population: The intention-to-treat (ITT) approach will be used for response to treatment data analysis of this trial.
Measure: Count of Participants; unit: Participants
Arm/Group | IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion/Time Point
Number analyzed (Participants) | 6
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 1
  Stable Disease (SD) | 2
  Progressive Disease (PD) | 3

ADVERSE EVENTS:
Time Frame: Day 0 to 28 days ± 7 business days from the last dose administered.
Arm/Group | IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion/Time Point
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion/Time Point (N=7)
Clostridial sepsis (Blood and lymphatic system disorders) | 1 — Multi-organ dysfunction syndrome and clostridial sepsis were experienced by the same patient leading to death. The principal investigator attributed these two SAEs as unlikely related to IFx-Hu2.0.
Multiple organ dysfunction syndrome (General disorders) | 1 — Multi-organ dysfunction syndrome and clostridial sepsis were experienced by the same patient leading to death. The principal investigator attributed these two SAEs as unlikely related to IFx-Hu2.0.
Pneumatosis (Gastrointestinal disorders) | 1 — The principal investigator attributed this SAE as unlikely related to IFx-Hu2.0.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion/Time Point (N=7)
Injection site reaction (General disorders) | 5
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Erythema (General disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Insomnia (Psychiatric disorders) | 2
Hypertension (Vascular disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Lymphedema (Vascular disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Moffitt shall be free to publish any academic articles, presentations, or abstracts of the Study results (including supporting data); provided that any such manuscript is first submitted to Company thirty (30) days prior to the proposed publication date so that Company may take any action necessary to protect its confidential information and intellectual property rights prior to said publication.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT03655756/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT03655756/ICF_001.pdf